CLINICAL TRIAL: NCT05638997
Title: Effects of Different Treatment Methods Applied to Spine in Chronic Non-Spesific Low Back Pain: A Randomized Controlled Trial
Brief Title: Effects of Different Treatment Methods Applied to Spine in Chronic Non-Spesific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Erkan Erol, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GaziosmanpasaU_Erol_01
Record Dates: First submitted 2022-11-16; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic Low Back Pain; Physiotherapy; Mulligan; Instrument Assisted Manipulation; Core Exercise
MeSH Terms: interventions — Movement

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Instrument Assisted Manipulation Group (Experimental): Instrument Assisted Manipulation + Core exercises
  Interventions: Other: Instrument assisted manipulation + Core exercises
- Mulligan Mobilization with Movement Group (Experimental): Mulligan Mobilization with Movement + Core exercises
  Interventions: Other: Mulligan mobilization with movement + Core exercises
- Control group (Active Comparator): Core exercises
  Interventions: Other: Core exercises

INTERVENTIONS:
Other: Instrument assisted manipulation + Core exercises — The effect of Instrument assisted manipulation on chronic non-spesific low back pain
  Arms: Instrument Assisted Manipulation Group
Other: Mulligan mobilization with movement + Core exercises — The effect of Mulligan mobilization with movement on chronic non-spesific low back pain
  Arms: Mulligan Mobilization with Movement Group
Other: Core exercises — The effect of core exercises on chronic non-spesific low back pain
  Arms: Control group

SUMMARY:
We aimed to investigate the effects of instrument assisted manipulation (IAM) and Mulligan mobilization with movement (MWM) on joint range of motion (ROM), pain, proprioception, endurance, back awareness and disability in individuals with chronic non-specific low back pain (CNSLBP). Fifthy one participants were randomly divided into 3 groups. The first was the Mulligan group, the second was the IAM group, and the third was the core exercise group. Visual Analogue Scale (VAS) was used to assess pain severity. Lumbal flexibility was evaluated with the fingertip-to-floor test. Oswestry disability index (ODI) and Roland Morris Disability Questionnaire (RMDQ) used to evaluate the disability. Fremantle back awareness questionnaire (FBAQ) used to evaluate back awareness. Joint ROM (lumbal flexion, lumbal extension and lumbal lateral flexion) and proprioception (30° lumbal flexion in standing, 30° lumbal flexion in sitting, 15° lumbal extension standing and lumbal neutral position) evaluated with JTECH digital dual inclinometer. McGill core endurance tests were used for core endurance assessment. McGill core endurance assessment consists of 3 tests. These: Flexor endurance test, lateral endurance test and extensor endurance test.

DETAILED DESCRIPTION:
IAM and Mulligan MWM interventions were applied 3 days a week for 2 weeks in total 6 sessions. All 3 groups did same core exercise program. The exercise program was done from the baseline for 6 weeks, 3 days a week, for a total of 18 sessions. Outcome measurements were done at baseline, at the end of the 2nd week, and at the end of the 6th week. The researcher who performed the outcome measurements did not know the participant's group. Assessment and treatment were performed by two different researchers with 8 years of professional experience. Visual Analogue Scale (VAS) was used to assess pain severity. Lumbal flexibility was evaluated with the fingertip-to-floor test. Oswestry disability index (ODI) and Roland Morris Disability Questionnaire (RMDQ) used to evaluate the disability. Fremantle back awareness questionnaire (FBAQ) used to evaluate back awareness. Joint ROM (lumbal flexion, lumbal extension and lumbal lateral flexion) and proprioception (30° lumbal flexion in standing, 30° lumbal flexion in sitting, 15° lumbal extension standing and lumbal neutral position) evaluated with JTECH digital dual inclinometer. The measurement of the joint ROM in the lumbal region with the dual inclinometer technique is a reliable method. McGill core endurance tests were used for core endurance assessment. McGill core endurance assessment consists of 3 tests. These: Flexor endurance test, lateral endurance test and extensor endurance test.

ELIGIBILITY:
Inclusion Criteria:

* LBP for at least 3 months
* Diagnosis of non-specific LBP
* 20-55 ages.

Exclusion Criteria:

* Red flag symptoms related to LBP
* Neurological findings
* Pain radiating to the leg
* Undergone spinal surgery
* Pathology of the spine (fracture, tumor, spondylolisthesis, spinal stenosis, cauda equina syndrome).

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline visual analogue scale at 2nd and 6th weeks | Baseline, 2nd week, 6th week
  Pain assessment. The minimum score of the visual analogue scale is 0, and the maximum score is 10. Higher scores indicate worse outcome.
Change from baseline fingertip-to-floor test at 2nd and 6th weeks | Baseline, 2nd week, 6th week
  Lumbal flexibility
Change from baseline joint ROM measurement with digital inclinometer at 2nd and 6th weeks | Baseline, 2nd week, 6th week
  Lumbal flexion, lumbal extension and lumbal lateral flexion
Change from baseline proprioception measurement with digital inclinometer at 2nd and 6th weeks | Baseline, 2nd week, 6th week
  30° lumbal flexion in standing, 30° lumbal flexion in sitting, 15° lumbal extension standing and lumbal neutral position
Change from baseline Oswestry disability index at 2nd and 6th weeks | Baseline, 2nd week, 6th week
  Disability assessment. The minimum score of the Oswestry disability index is 0, and the maximum score is 50. Higher scores indicate worse outcome.
Change from baseline Roland Morris disability questionnaire at 2nd and 6th weeks | Baseline, 2nd week, 6th week
  Disability assessment. The minimum score of the Roland Morris disability questionnaire is 0, and the maximum score is 24. Higher scores indicate worse outcome.
Change from baseline Fremantle back awareness questionnaire at 2nd and 6th weeks | Baseline, 2nd week, 6th week
  Back awareness assessment. The minimum score of the Fremantle back awareness questionnaire is 0, and the maximum score is 36. Higher scores indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Erkan Erol, PhD, Principal Investigator — Tokat Gaziosmanpaşa University
Locations (1):
- Faculty of Health Sciences, Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No